CLINICAL TRIAL: NCT06130579
Title: Interferon-α for Preventing Relapse in TP53+ Myeloid Malignancy Post Allo-HSCT
Brief Title: Interferon-α for TP53 Myeloid Malignancy Post Allo-HSCT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Xiao-Jun Huang, Professor, Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IFN-α for preventing relapse
Record Dates: First submitted 2023-11-08; First posted 2023-11-14 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-03

CONDITIONS: Myeloid Leukemia; Myelodysplastic Syndromes
Keywords: IFN-α; Preventing relapse; allo-HSCT
MeSH Terms: conditions — Leukemia, Myeloid; Myelodysplastic Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- IFN-α application in TP53+ myeloid malignancy (Experimental)
  Interventions: Drug: IFN-Α

INTERVENTIONS:
Drug: IFN-Α — Leukemia-associated immunophenotyping (LAIPs) was performed by flow cytometry at +1 month and +2 month after HSCT. If MRD was negative on two consecutive flow cytometry assays, interferon-α prophylaxis was initiated on day +75 after transplantation, and cyclosporine was tapered on day +100 after transplantation. The dose of interferon-α was 3 million units/time, subcutaneously injected twice a week. Cycles were given every 4 weeks until hematologic relapse or up to 6 cycles.

SUMMARY:
To investigate the efficacy of interferon-α prophylaxis in patients with acute myeloid leukemia (AML) and myelodysplastic syndrome (MDS) with TP53 mutation who were negative for minimal residual disease (MRD) by flow cytometry within 2 months after allogeneic hematopoietic stem cell transplantation. To explore the efficacy of interferon-α in reducing the relapse rate of AML/MDS patients with TP53 mutation after allogeneic hematopoietic stem cell transplantation (allo-HSCT).

ELIGIBILITY:
Inclusion Criteria:

1. Myelodysplastic syndrome (MDS) diagnosed according to the 2022 International Consensus Classification of Myeloid Neoplasms and Acute Leukemia (2022ICC) criteria, acute myeloid leukemia (AML) with TP53 mutation (unrestricted remission status), minimal residual disease (MRD) monitored by flow cytometry within 2 months after receiving the first allogeneic hematopoietic stem cell transplantation Negative patients
2. Male or female, aged 12-65 years
3. Karnofsky score >60, estimated survival time >3 months
4. No history of severe graft-versus-host disease (GVHD), uncontrolled GVHD, or severe systemic organ dysfunction:

   1. Absolute neutrophil count (ANC) greater than 0.5×109/L
   2. Creatinine < 1.5mg/dL
   3. Cardiac ejection index >55%
5. Signed informed consent.

Exclusion Criteria:

1. severe cardiac, renal, or liver dysfunction
2. combined with other malignant tumors requiring treatment
3. inability to understand or adhere to the study protocol due to clinical symptoms of brain dysfunction or severe mental illness
4. patients who are unable to complete the necessary treatment plan and follow-up observation
5. patients with severe acute anaphylaxis
6. clinically uncontrolled severe life-threatening infections
7. patients enrolled in other clinical trials
8. other reasons considered by the investigator to be inappropriate for clinical trial participants.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
The incidence of relapse | 1 year post HSCT
  Disease relapse was defined as blasts ≥ 5% post transplantation.

SECONDARY OUTCOMES:
The incidence of positive minimal residual disease post allo-HSCT | 1 year post HSCT
  Positive MRD was defined as leukemia-associated immunophenotyping (LAIPs) by flow cytometry.
The incidence of acute and chronic graft versus host disease (GvHD) | aGvHD within 100 days and cCvHD within 1 year
  The severity of acute GvHD (aGvHD) and chronic GvHD (cGvHD) was evaluated according to standard criteria.
The incidence of non-relapse mortality | 1 year post HSCT.
  The incidence of non-relapse mortality
The probability of progression free survival | 1 year post HSCT.
  Survival without disease progression
The probability of overall survival (OS) | 1 year post HSCT.
  OS was defined as the time from transplantation to death from any cause or to the last follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Deparment of Hematology, Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No